CLINICAL TRIAL: NCT03397641
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Serial Cohort Dose-Escalation Study of Intravenously Administered HBI-3000
Brief Title: A Phase 1 Study of HBI-3000
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBI-3000-301; 2017-003642-24 (EudraCT Number)
Record Dates: First submitted 2017-11-28; First posted 2018-01-12 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — sulcardine sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): x mg HBI-3000 as x mL of a 50 mg/mL solution for intravenous infusion. Doses of HBI-3000 (Cohorts A to G) may range from 20 mg to a level at which it is expected that the drug exposure will not exceed an AUC(0-t) of 20 µg.h/mL and Cmax of 20 µg/mL (based on the NOAEL) in both 14-day repeat-dose toxicology species rat and minipig) and the expected therapeutic dose.
  Interventions: Drug: HBI-3000
- Placebo (Placebo Comparator): Matching placebo for x mg HBI-3000 as x mL of a 50 mg/mL solution for intravenous infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HBI-3000 — Small molecule, multi-ion channel blocker
  Other Names: Sulcardine sulfate
  Arms: Active
Other: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
This is a Phase 1 randomised, double-blind, placebo-controlled, serial cohort, dose-escalation study in healthy adult volunteers. It is planned to enroll 5 cohorts (Cohorts A to E) of 8 subjects. Up to 2 additional cohorts (Cohorts F and G) may be enrolled as needed to establish the safety profile of HBI-3000 over a clinically relevant range of doses. Subjects will be randomly assigned to receive a single dose of HBI-3000 or matching placebo in a sequential escalating manner (Regimens A to E and optional Regimens F and G), with a minimum of 7 days and a maximum based on logistics of interim review between dose groups.

As a safety precaution, in each cohort a sentinel dosing group of n = 2 (1 active:1 placebo) will be dosed at least 24 h ahead of the main group. Safety and tolerability will be assessed by the principal investigator or medically-qualified designee before continuing with dosing the remaining subjects. The first 2 subjects will be allocated to active or placebo in a 1:1 ratio. The remaining 6 subjects will be allocated to active or placebo in a 5:1 ratio.

Doses of HBI-3000 may range from 20 mg to a level at which it is expected that the drug exposure will not exceed an AUC(0-t) of 20 μg.h/mL and Cmax of 20 μg/mL (based on the no-observed-adverse-effect levels [NOAEL] in both 14 day repeat dose toxicology species the rat and minipig) and the expected therapeutic dose range. Following administration to each cohort, there will be an interim data review during which the PK and safety data will be reviewed to determine the dose to be administered in the next cohort. Dose escalation for serial cohorts will progress unless safety concerns preclude further dose escalation. If the selected dose does not provide the required data, a previously tested dose may be used in a subsequent cohort. However, if the dose level met the dose escalation stopping criteria, that dose level must not be repeated. A previously untested intermediate dose may also be used in a subsequent cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Age 18 to 50 years
3. Body mass index of 18.0 to 30.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Minimum body weight of 60 kg
5. Must be willing and able to communicate and participate in the whole study
6. Normal hepatic function as evidenced by AST and alanine aminotransferase (ALT) <1.5 × ULN and alkaline phosphatase (ALP) and total bilirubin within the normal range
7. Haemodynamically stable with systolic BP 90 to 150 mm Hg, diastolic BP <95 mmHg and resting HR ≥45 and ≤100 bpm
8. Forced expiratory volume in 1 s (FEV1) >80% predicted value and FEV1/ forced vital capacity (FVC) ratio >0.7
9. Must provide written informed consent
10. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study.
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
7. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
8. Females of childbearing potential who are pregnant or lactating (all female subjects must have a negative pregnancy test). A woman is considered of childbearing potential unless she is permanently sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy) or is postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle-stimulating hormone [FSH] concentration ≥40 IU/L)
9. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
10. Clinically significant abnormal biochemistry, haematology, coagulation or urinalysis as judged by the investigator, including:

    * Serum K <3.5 mmol/L
    * Serum magnesium concentration of <0.7 mmol/L
    * Serum phosphate <2.5 or >4.5 mg/dL
11. Positive drugs of abuse test result
12. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
13. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <80 mL/min using the Cockcroft-Gault equation
14. Evidence of any clinically relevant acute or chronic medical illness, including renal, hepatic, haematological, endocrine, pulmonary (including asthma), oncologic, neurologic or gastrointestinal disease, or psychiatric disorder, as judged by the investigator
15. History or presence of clinically significant cardiovascular disease, including coronary artery disease, myocardial infarction or ischemia, congestive heart failure, valvular disease, congenital heart disease or prior cardiac surgery
16. History or presence of cardiac arrhythmia or conduction abnormalities, including long-QT syndrome, TdeP, Wolff-Parkinson-White syndrome or bradycardia (<45 bpm)
17. QTcF interval >450 or QRS >120 msec
18. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
19. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
20. Donation or loss of greater than 400 mL of blood within the previous 3 months
21. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol and HRT/hormonal contraception) or herbal remedies in the 14 days before IMP administration (see Section 11.4). Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
22. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Physical Examination (Safety and Tolerability) | Change from screening (3 to 28 d prior to dosing), admission (2 d prior to dosing), 48 h post-start of infusion, and 7 d +/- 1 d post-start of infusion (follow-up visit)
  Typical physical examination, including general appearance; head, neck, and thyroid; ears, nose, and throat; cardiovascular; respiratory; lymph nodes; abdomen; dermatological; musculoskeletal; neurological/CNS; ocular/ophthalmology; and other (as specified) evaluation
Safety Labs (Safety and Tolerability) | Change from screening (3 to 28 d prior to dosing), 1 d prior to dosing, 24 h and 48 h post-start of infusion, and 7 d +/- 1 d post-start of infusion (follow-up visit)
  Hematology (hemoglobin[g/L], HCT[%], RBC[x10^12/L], MCV[fL], MCH[pg], MCHC[g/L], platelet[x10^9/L], WBC[x10^9/L], neutrophils[x10^9/L], lymphocytes[x10^9/L], monocytes[x10^9/L], eosinophils[x10^9/L], basophils[x10^9/L], hematocrit[%]), coagulation (prothrombin time[s], APTT[s]), clinical chemistry (Na[mmol/L], K[mmol/L], Cl[mmol/L], bicarbonate[mmol/L], urea[mmol/L], creatinine[µmol/L], bilirubin[µmol/L], direct conj bilirubin[µmol/L], alkaline phosphatase[IU/L], aspartate aminotransferase[IU/L], alanine aminotransferase[IU/L], creatinine kinase[IU/L], gamma glutamyl transferase[IU/L], total protein[g/L], albumin[g/L], Ca[mmol/L], Mg[mmol/L], P[mmol/L], uric acid[µmol/L], random blood glucose[mmol/L], fasting blood glucose[mmol/L], triglycerides[mmol/L], fasting triglycerides[mmol/L], creatinine clearance[mL/min]), virology (Hepatitis B surface[+/-], Antigen[+/-], Hepatitis C[+/-], Antibody[+/-], HIV Antibody[+/-]); and FSH(IU/L) and beta H.C.G. serum(+/-)
Urinalysis (Safety and Tolerability) | Change from screening (3 to 28 d prior to dosing), admission (2 d prior to dosing), 24 h and 48 h post-start of infusion, and 7 d +/- 1 d post-start of infusion (follow-up visit)
  Bilirubin (-/+; +, ++, +++), urobilinogen (-/+; 2, 4, 8, 12 mg/dL), ketones (-/+; trace, +, ++, +++), glucose (-/+; 50, 100, 250, 500, ≥1000 mg/dL), pH (5.0, 6.0, 6.5, 7.0, 8.0, 9.0), hCG (female subjects; -/+), specific gravity (1.000, 1.005, 1.010, 1.015, 1.020, 1.025, 1.030), protein (-/+; trace, 30, 100, 500 mg/dL), blood (-/+; +ca.5-10, ++ca.50, +++ca.300, ca.5-10, ca.50, ca.300 ery/µL), nitrites (-/+; light pink, dark pink), leukocytes (-/+; ca.25, ca.75, ca.500 leuko/µL) (performed using dipsticks; if positive, tick correct result), microbiology (WBS [HPF], RBCS [HPF], hyaline casts [HPF], granular casts [HPF], cellular casts [HPF]) and urine microscopy (both at the discretion of the investigator based on urinalysis results), and drugs of abuse (amphetamines [+/-], barbiturates [+/-], benzodiazepines [+/-], cocaine [+/-], marijuana/cannabis [+/-], methadone [+/-], methamphetamine/ecstasy [+/-], morphine/opiates [+/-], phencyclidine [+/-], tricyclic antidepressants [+/-])
Pulmonary Function Tests (Safety and Tolerability) | Change from screening (3 to 28 d prior to dosing), pre-dose (within 24 h prior to dosing), and 0.75 h and 4 h post-start of infusion
  The following lung function tests will be performed using a standard calibrated spirometer: FEV1 (L), FVC (L), peak expiratory flow rate (PEFR) (L/min), and FEV1/FVC (%)
12-Lead ECG (Safety and Tolerability) | Change from screening (3 to 28 d prior to dosing), admission (2 d prior to dosing), pre-dose (within 24 h prior to dosing), 0.25 h, immediately prior to end of infusion, 1, 4, 6, 12, 24, and 48 h, and 7 d +/- 1 d post-start of infusion
  Measured after subject has been in supine position for at least 5 min.
Holter ECG (Safety and Tolerability) | Data extractions on Day -1 will be time matched to the planned time of dosing on Day 1 (i.e., 12 extractions); the extraction time points on Day 1 are: pre-dose, 0.25 h, 0.5 h, 0.75 h, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 24 h post-start of infusion
  Continuous ECG monitoring; subjects to be in supine position for at least 0.25 h before each extraction
Telemetry ECG (Safety and Tolerability) | To commence approximately 10 min before dosing up to 6 h post-start of infusion
  No data are collected (safety monitoring); if cardiac monitoring shows a potentially significant abnormality, a clinical assessment of the subject will be performed, including a 12-lead ECG, and treatment given.
Vital Signs (Safety and Tolerability) | Change from screening (3 to 28 d prior to dosing), admission (2 d prior to dosing), pre-dose (within 24 h prior to dosing), 0.25 h, immediately prior to end of infusion, 1, 2, 4, 6, 8, 12, 16, 24, 30, 36, and 48 h, and 7 d +/- 1 d post-start of infusion
  Blood pressure (mmHg), heart rate (bpm), oral temperature (degrees C or degrees F)
Adverse Events (Safety and Tolerability) | 0.25 h post-start of infusion through 7 d +/- 1 d post-start of infusion (follow-up visit)
  All AEs are documented, including the date and time of onset, a description of the AE, severity, duration, actions taken, outcome and investigator's current opinion on the relationship between HBI-3000 and the event.

SECONDARY OUTCOMES:
HBI-3000 Levels Over Time in Plasma (Cmax) | Change in Cmax from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Peak Plasma Concentration, Cmax (µg/mL)
HBI-3000 Levels Over Time in Plasma (Tmax) | Change in Tmax from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Time to Reach the Peak Plasma Concentration, Tmax (h)
HBI-3000 Levels Over Time in Plasma (AUC(0-last)) | Change in AUC(0-last) from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Area Under the Plasma Concentration versus Time Curve from Time Zero to Time of Last Measurable Concentration, AUC(0-last) (µg·h/mL)
HBI-3000 Levels Over Time in Plasma (AUC(0-inf)) | Change in AUC(0-inf) from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Area Under the Plasma Concentration versus Time Curve from Time Zero to Infinity, AUC(0-inf) (µg·h/mL)
HBI-3000 Levels Over Time in Plasma (AUC(0-24h)) | Change in AUC(0-24h) from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Area Under the Plasma Concentration versus Time Curve from Time Zero to Time 24h, AUC(0-24h) (µg·h/mL)
HBI-3000 Levels Over Time in Plasma (AUC%extrap) | Change in AUC%extrap from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Area Under the Plasma Concentration versus Time Curve Extrapolated from Time t to Infinity as a Percentage of total AUC, AUC%extrap (%)
HBI-3000 Levels Over Time in Plasma (lambda-z) | Change in lambda-z from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Terminal Disposition Rate Constant/Terminal Rate Constant, lambda-z (1/h)
HBI-3000 Levels Over Time in Plasma (T1/2) | Change in T1/2 from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Elimination Half Life, T1/2 (h)
HBI-3000 Levels Over Time in Plasma (CL) | Change in CL from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Apparent Total Clearance of the Drug from Plasma, CL (mL/h·kg)
HBI-3000 Levels Over Time in Plasma (CLr) | Change in CLr from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Renal Clearance of the Drug from Plasma, CLr (mL/h·kg)
HBI-3000 Levels Over Time in Plasma (Vz) | Change in Vz from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Apparent Volume of Distribution during Terminal Phase, Vz (L/kg)
HBI-3000 Levels Over Time in Plasma (Vss) | Change in Vss from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Apparent Volume of Distribution at Steady State, Vss (L/kg)
HBI-3000 Levels Over Time in Plasma (MRT) | Change in MRT from pre-dose (within 24 h prior to dosing), and 0.25 h, immediately prior to end of infusion, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 16 h, 24 h, 30 h, 36 h, 48 h, 72 h post-start of infusion
  Mean Residence Time, MRT (h)
HBI-3000 Levels Over Time in Urine (Ae) | Change in Ae from pre-dose (within 24 h prior to dosing), and 0-6 h, 6-12 h, 12-24 h post-start of infusion
  Amount of Unchanged Drug Excreted into the Urine, Ae (µg)
HBI-3000 Levels Over Time in Urine (CumAe) | Change in CumAe from pre-dose (within 24 h prior to dosing), and 0-6 h, 6-12 h, 12-24 h post-start of infusion
  Cumulative Recovery of Unchanged Drug Excreted into the Urine, CumAe (µg)
HBI-3000 Levels Over Time in Urine (%Ae) | Change in %Ae from pre-dose (within 24 h prior to dosing), and 0-6 h, 6-12 h, 12-24 h post-start of infusion
  Amount of Unchanged Drug Excreted into the Urine as a Percentage of the Administered Dose, %Ae (%)
HBI-3000 Levels Over Time in Urine (Cum%Ae) | Change in Cum%Ae from pre-dose (within 24 h prior to dosing), and 0-6 h, 6-12 h, 12-24 h post-start of infusion
  Cumulative Recovery of Unchanged Drug Excreted into the Urine as a Percentage of the Dose, Cum%Ae (%)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, Study Director — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided